CLINICAL TRIAL: NCT01023932
Title: Cochlear Implants in Children With Auditory Neuropathy/ Auditory Dys-Synchrony
Brief Title: Auditory Neuropathy and Cochlear Implants
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Ana Claudia Martinho de Carvalho
Other Study IDs: NADA2009
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Cochlear Implants; Auditory Neuropathy
MeSH Terms: conditions — Auditory neuropathy | interventions — Cochlear Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Auditory Neuropathy Patients
  Interventions: Device: Cochlear Implants

INTERVENTIONS:
Device: Cochlear Implants

SUMMARY:
The electrical stimulation generated by the Cochlear Implant (CI) may improve the neural synchrony and hence contribute to the development of auditory skills in patients with Auditory Neuropathy / Auditory Dys-synchrony (AN/AD). Goal: The goal of the research was to evaluate the auditory performance and the characteristics of the electrically evoked compound action potential (ECAP) in a group of 18 cochlear implants recipients with AN/AD.The auditory perception was evaluated by sound field thresholds and speech perception tests. To evaluate ECAP's characteristics, the threshold and amplitude of neural response together with the amplitude growth and recovery functions were evaluated at 80Hz stimulation rate.The CI was seen as an efficient resource to develop auditory skills in 94% of the AN/AD patients considered by the research. The auditory perception benefits as well as the possibility to measure the ECAP showed that the electrical stimulation could compensate the neural dys-synchrony caused by the AN/AD. However, a unique clinical procedure cannot be proposed at this point. Therefore, a careful and complete evaluation of each AN/AD patient before recommending the Cochlear Implant is advised

ELIGIBILITY:
Inclusion Criteria:

* All children with AN/AD who had received the cochlear implant during the research´s period.

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Children with auditory neuropathy who had received a cochlear implant
Sampling Method: Non-Probability Sample
Dates: Start 2006-09; Study Completion 2009-09

PRIMARY OUTCOMES:
The CI was seen as an efficient resource to develop auditory skills in 94% of the AN/AD patients considered by the research.

CONTACTS AND LOCATIONS:
Locations (1):
- Bionic Ear Center, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] de Carvalho ACM, Bevilacqua MC, Sameshima K, Filho OAC. Auditory neuropathy/Auditory dyssynchrony in children with Cochlear Implants. Braz J Otorhinolaryngol. 2011 Jul-Aug;77(4):481-487. doi: 10.1590/S1808-86942011000400012. PMID 21860975